CLINICAL TRIAL: NCT01810107
Title: Study to Evaluate the Efficacy of Optical Imaging to Evaluate the Anatomy of the Developing Pediatric Vocal Fold
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Christopher Hartnick, M.D., Principal Investigator, Massachusetts Eye and Ear Infirmary
Other Study IDs: 11-006H
Record Dates: First submitted 2012-10-19; First posted 2013-03-13 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Vocal Fold Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children Examined with the OCT Probe: Children undergoing surgery will also have the Optical Coherence Tomography probe.
  Interventions: Procedure: Children Examined with the OCT Probe
- Adults: Adults undergoing surgery will also have the Optical Coherence Tomography probe.
  Interventions: Procedure: Children Examined with the OCT Probe

INTERVENTIONS:
Procedure: Children Examined with the OCT Probe — The child undergoing therapy will have the Optical Coherence Tomography (OCT) probe to examine the vocal fold.

SUMMARY:
The specific aim of this study is to develop a growth and development chart (similar to a height or weight chart for children) that identifies the pattern of development of the pediatric vocal cord lamina propria from a single to a three layer structure. A secondary aim is to identify whether this growth chart shows a pattern of linear development or whether there are clear critical periods of development.

DETAILED DESCRIPTION:
The goal of this study is to identify critical periods of development when the lamina propria structure of the pediatric vocal fold matures. A Universal Modular Glottiscope will be utilized for adequate laryngeal exposure. An operating microscope will be used for magnification. This setup will allow for the Optical Coherence Tomography (OCT) imaging probe to be introduced using a laryngoscope to provide stability. The optical imaging probe will then be directed, or gently applied towards, the glottal surface, and an image field of 500 microns x 500 microns x 350 microns will be obtained. As the probe is moved along the medial and superior mucosal surfaces of the vocal folds, "real-time" images will be obtained and digitally stored for review. The digitally stored images will be assessed and analyzed for their optical characteristics. The optical imaging probe will then be withdrawn from the patient and the original operative procedure will then be performed. Images can be attained in both "non-contact" mode (where the probe tip remains in the space between each vocal fold) and "contact" mode (where the probe tip is gently placed against the glottal tissue to compress it). The contact mode allows for deeper imaging (much like an ultrasound), which would be useful in situations involving larger (thicker) vocal folds. The study will end when images are acquired from a range of developmental ages to be able to refine the optical characteristics of the optical imaging system.

Adults have also been included in this study for comparison as OCT imaging in adults may confirm the number of vocal fold layers compared to children.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1 month to 18 (and adults >18) undergoing laryngoscopy and bronchoscopy for airway evaluation where the patients will be already scheduled for general anesthesia with intravenous catheter placement as part of standard routine.
* Children (and adults) undergoing any otolaryngology procedure where there is no indication of airway obstruction or risk of abnormal vocal chords. For instance, children undergoing adenoidectomy, sinus surgery or tracheotomy are all good candidates for studying the normal vocal chord development.
* Children whose parents have given and signed an informed consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization and who have signed an assent form (if they are 7 and older) agreeing to participate in the study. Eligibility will be determined by the Principal Investigator.
* Adults who have given and signed an informed consent and HIPAA Authorization.

Exclusion Criteria:

* Children (or adults) with any form of laryngeal anomaly or pathology.
* Children who have previously been intubated.
* Children, adolescents, and adults who smoke. Exclusion will be determined by the Principal Investigator.

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children ages 1 month to 18 (and adults >18) undergoing laryngoscopy and bronchoscopy for airway evaluation where the patients will be already scheduled for general anesthesia with intravenous catheter placement as part of standard routine.
Sampling Method: Non-Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Vocal Fold Development | 30 seconds to a minute, in the operating room, before the otolaryngology procedure that they are originally there for. This time frame is all that is needed to image their vocal cords.
  The goal of this study is to identify critical periods of development when the lamina propria structure of the pediatric vocal fold matures. The major analysis will be to validate the age dependent laminar structure using a cohort of 720 subjects between age 0-18 as well as estimate the probability of future events of developing two- or three laminar structure given a subject's age. We will perform one-sided two-sample binomial tests to examine as well as model the patterns of the rates of bi- and tri-laminar structure patterns by using logistic model or discrete or continuous time Cox's proportional hazards model of which the predictor variables are determined based on the discriminant model described above. In addition, as a parallel approach we will analyze the Optical Coherence Tomography (OCT) data of each of the trilaminar system by using linear or curve-linear regression models which will provide a prediction model of the mean OCT at various critical ages.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No